CLINICAL TRIAL: NCT01593072
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Dose-Escalation A Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Dose-Escalation Study to Assess the Safety, Tolerability and Pharmacokinetics of AVI-7537 in Healthy Adult Volunteers
Brief Title: A Study to Assess the Safety, Tolerability and Pharmacokinetics of AVI-7537 in Healthy Adult Volunteers
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated for convenience of the Government due to funding constraits
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7537-us-101; W9113M-10-C-0056 (Other Grant/Funding Number: Transformational Medical Technologies, US Dept. of Defense)
Record Dates: First submitted 2012-05-03; First posted 2012-05-07 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Ebola Hemorrhagic Fever
Keywords: Multiple Ascending Dose (MAD); Ebola Virus; Post Exposure Prophylaxis; EHF
MeSH Terms: conditions — Hemorrhagic Fever, Ebola | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AVI-7537 (Active Comparator): AVI-7537
  Interventions: Drug: AVI-7537
- Placebo (Other): Normal Saline Solution (NSS)
  Interventions: Other: Normal Saline Solution (NSS)

INTERVENTIONS:
Drug: AVI-7537 — Cohort 1: AVI-7537 at 4.5 mg/kg IV; Cohort 2: AVI-7537 at 9 mg/kg IV;Cohort 3: AVI-7537 at 15 mg/kg IV; Cohort 4: AVI-7537 at 30 mg/kg IV
  The amount of AVI-7537 required to administer the required dose will be diluted to a volume of approximately 150 mL with normal saline solution (NSS) and given by IV infusion over 30 minutes once a day for 14 days. Infusions will be administered at approximately the same time each day.
  Arms: AVI-7537
Other: Normal Saline Solution (NSS) — Normal Saline Solution (NSS)
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of healthy male and female subjects with intravenous (IV) infusions of AVI 7537 compared to matched placebo in and to evaluate the pharmacokinetics (PK).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and tolerability of 14 once daily intravenous (IV) infusions of ascending doses of AVI 7537 compared to matched placebo in healthy male and female subjects.

To evaluate the pharmacokinetics (PK) of 14 once daily doses of AVI-7537 in healthy male and female subjects

ELIGIBILITY:
Inclusion Criteria:

A subject must meet all of the following criteria to be eligible for this study.

1. Man or woman 18 to 50 years of age, inclusive, at the time of screening.
2. Body mass index 18 kg/m2 to 35 kg/m2, inclusive, at the time of screening and Check-in (Day -1).
3. Good general health (no chronic health conditions) as determined by the Investigator.
4. Female subjects must be of non-childbearing potential (e.g., be confirmed post-menopausal or have undergone surgical sterilization) or must, in conjunction with their sexual partner(s), use 2 forms of medically acceptable contraception (e.g., oral contraception in conjunction with a male condom) during the screening period and for the entire duration of the study including the 28-day post last dose follow-up.
5. Male subjects must either be sterile or agree to use, for the entire duration of the study including the 28 day post last dose follow-up, a male condom and the female sexual partner must also use a medically acceptable form of birth control (e.g. oral contraceptives).
6. Male subjects must agree to not donate sperm for at least 30 days after the last infusion of study medication.
7. Able to understand the requirements of the study, to provide written informed consent (as evidenced by signature on an informed consent document that is approved by an Institutional Review Board [IRB]), and agreeable to abiding by the study restrictions.

Exclusion Criteria:

A subject who meets any of the following criteria will be excluded from this study.

1. Pregnancy or breastfeeding.
2. A positive urine or blood screen for drugs of abuse, including alcohol.
3. Use of any tobacco- or nicotine-containing products (including but not limited to cigarettes, pipes, cigars, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to Check-in (Day -1).
4. A positive cotinine test indicating recent nicotine use.
5. Donated blood within 90 days or plasma within 30 days of first dose on Day 1.
6. Active substance abuse or any medical or psychiatric condition that could jeopardize the subject's safety or the subject's ability to comply with the protocol.
7. Use of any medications apart from vitamins, acetaminophen, or hormonal contraception within 14 days of first dose on Day 1. Subjects with mild seasonal allergies may use antihistamines at the discretion of the Investigator after approval by the Sponsor Medical Monitor.
8. Participation in any interventional clinical trial within 45 days of first dose on Day 1 (i.e., received any other investigational drug).
9. Recipient of an organ transplant (solid or hematopoietic).
10. Prolonged QTcF interval > 440 ms for males or > 460 ms for females using the average of the triplicate electrocardiograms (ECGs) collected during screening, on Day -1, or just prior to dosing on Day 1.
11. Other clinically significant ECG abnormality, as determined by the Investigator.
12. Any clinically significant abnormal hematology, chemistry, coagulation, or urinalysis value, as determined by the Investigator.
13. Glomerular filtration rate (GFR) of < 80 mL/min, based on the Modification of Diet in Renal Disease equation.
14. Urine-albumin-to-creatinine ratio (UACR) > 30 mg/g.
15. Positive test for human immunodeficiency virus (HIV-1 serology) or known HIV infection.
16. Positive result for hepatitis B surface antigen (HBsAg) or for hepatitis C virus (HCV) antibody.
17. Use of alcohol-containing foods or beverages within 72 hours prior to Check-in on Day -1.
18. Use of caffeine-containing foods or beverages within 24 hours prior to Check-in on Day -1.
19. Febrile illness or significant infection within 48 hours before administration of the first dose of study drug on Day 1.

Note: Inclusion of each subject will be reviewed with a member of AVI BioPharma Clinical Personnel prior to enrollment in the trial. Written approval from a member of AVI BioPharma Clinical Personnel is required prior to randomization.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
The outcome measures are Serial PK Day 1 over 24 hrs(pre-dose,10 min post,30 min post, 1hr 1.5,2,4,6, 8, 12,16,24,28,32,36, and 48 hrs post-dose), daily through level and on Day 14 (last day of dosing) serial PK until 48 hrs post last dose. | 2 weeks
  The outcome measures are Serial PK Day 1 over 24 hours (pre-dose, 10 minutes post-dose , 30 minutes, 1 hour, 1.5, 2, 4, 6,. 8, 12,16,24 hours post-dose), daily trough level and on Day 14 (last day of dosing). PK Day 14 over 48 hours (post-dose, 10 minutes, 1.5, 2, 4, 6, 8, 12, 16, 24, 28, 32, 36, and 48 hours post-dose (collection of plasma pre-dose on Day 14 will also serve as the trough sample for that day).

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of 14 once daily doses of AVI-7537 in healthy male and female subjects, | 2 weeks
  Efficacy will not be assessed in a Phase I study.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Heald, MD, Principal Investigator — Sarepta Therapeutics, Inc.
Locations (1):
- Quintiles Phase I Services, Overland Park, Kansas, United States